CLINICAL TRIAL: NCT00212680
Title: Controlled Study of ONO-1101 in Patients With Postoperative Tachyarrhythmias in Japan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Organization: Ono Pharmaceutical Co. Ltd (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-1101-1906
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Postoperative Supraventricular Tachyarrythmia
Keywords: ONO-1101,Landiolol Hydrochloride, Postoperative, Supraventricular Tachyarrhythmia
MeSH Terms: interventions — landiolol

INTERVENTIONS:
Drug: ONO-1101

SUMMARY:
The purpose of this study was to evaluate the dose-dependent effects of ONO-1101 on efficacy and safety in patients with postoperative supraventricular tachyarrhythmias.

ELIGIBILITY:
Inclusion Criteria:

1. 20-80 years old
2. Postoperative supraventricular tachyarrhythmias (sinus tachycardia, those with a heart rate of 120 beats/min or higher, and supraventricular arrhythmia, those with a heart rate of 100 beats/min or higher)
3. Within 7 days postoperatively
4. Other inclusion criteria as specified in the protocol

Exclusion Criteria:

1. Acute myocardial infarction (within 1 month after onset)
2. Severe heart failure (New York Heart Association functional class III or higher)
3. Atrioventricular block (grade II or higher),or sick sinus syndrome
4. Other exclusion criteria as specified in the protocol

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 1996-12; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving 20% reduction in heart rate at each dose

SECONDARY OUTCOMES:
Heart Rate, Blood pressure and 12-lead ECG

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Development Planning, Study Director — Ono Pharmaceutical Co. Ltd